CLINICAL TRIAL: NCT04015752
Title: Sepsis in Intensive Care Unit :Causes and Outcomes of Sepsis in Diabetics Versus Non Diabetics in Assiut University Hospital
Brief Title: Sepsis in ICU:Causes and Outcomes of Sepsis in Diabetics Versus Non Diabetics in Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Srour, Principle Investigator, Assiut University
Other Study IDs: Sepsis in ICU.
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Sepsis; Septic Shock
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Blood Gas Analysis; Kidney Function Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- diabetics: 1. Full history with special attention to:
     Causes of admission to ICU . Duration of DM when present, medication used, controlled or not.
  2. Complete physical examination with special attention to :
     Vital signs ( MAP, pulse, temp, RR). Signs of shock (cold clammy skin , oliguria, altered mental status ) Consciousness level. Source of infection (chest , abdomen ,catheter, JV canula,..).
  3. Laboratory investigations includes :
  CBC , Liver and kidney functions → baseline and follow up. Arterial Blood Gases (ABG). Lactic acid level. HBA1C. ESR, CRP →baseline and follow up.
  Culture :
  On admission Urine and blood as well as sputum culture acc. To the cause of infection. Culture from suspected site of infection in catheter related infections.
  Interventions: Diagnostic Test: culture from infected site
- non diabetics: 1. Full history with special attention to:
     Causes of admission to ICU . Duration of DM when present medication used, controlled or not.
  2. Complete physical examination with special attention to :
     Vital signs ( MAP, pulse, temp, RR) Signs of shock (cold clammy skin , oliguria, altered mental status ) Consciousness level. Source of infection (chest , abdomen ,catheter, JV canula,..).
  3. Laboratory investigations CBC , Liver and kidney functions → baseline and follow up HBA1C. ESR, CRP →baseline and follow up.
  Culture :
  On admission Urine and blood as well as sputum culture acc. To the cause of infection. Culture from suspected site of infection in catheter related infections.
  Interventions: Diagnostic Test: culture from infected site
- patients devoloped hyperglycemia in ICU only: Full history with special attention to:
  Causes of admission to ICU . Duration of DM when present medication used, controlled or not. 2. Complete physical examination with special attention to : Vital signs ( MAP, pulse, temp, RR) Signs of shock (cold clammy skin , oliguria, altered mental status ) Consciousness level. Source of infection (chest , abdomen ,catheter, CVP,..). 3. Laboratory investigations CBC , Liver and kidney functions → baseline and follow up HBA1C. ESR, CRP →baseline and follow up.
  Culture :
  On admission Urine and blood as well as sputum culture acc. To the cause of infection. Culture from suspected site of infection in catheter related infections.
  Interventions: Diagnostic Test: culture from infected site

INTERVENTIONS:
Diagnostic Test: culture from infected site — ESR ,CRP,CBC, Renal and Liver function will be done on admission and follow up Culture: On admission Urine and blood as well as sputum culture acc. To the cause of infection. Culture from suspected site of infection in catheter related infections.
  Other Names: HbA1C; Arterial Blood Gases; Lactic acid level; CBC; ESR; CRP; liver and kidney function tests

SUMMARY:
Clarify different causes of sepsis in patients admitted to ICU . as well asCompare causes and outcomes of sepsis between diabetics versus non diabetics .

3.Screening for the commonest organism causing sepsis in critically ill patients.

Determine better protocol therapy that help in decreasing mortality and morbidity in patients with sepsis in ICU.

DETAILED DESCRIPTION:
Sepsis is a physiologic, pathologic, and biochemical abnormalities induced by infection.

sepsis is considered as a leading cause of mortality and critical illness worldwide by many conservative estimates.

sepsis epidemiology studies worldwide revealed a highly variable incidence of 13-300 per 100,000 inhabitants per year for severe sepsis and 11 per 100,000 inhabitants per year for septic shock .

factors such as advancing age, immunosuppression and multi-drug-resistant infection play a role in increasing incidence of sepsis during recent decades .

patients who survive sepsis often have long-term physical, psychological, and cognitive disabilities with significant health and social implications.

Patients with diabetes mellitus have an increased risk of developing infections and sepsis and they constitute 20.1-22.7% of all sepsis patients.

Infection also remains an important cause of death in diabetics. The prevalence of diabetes mellitus in Intensive Care Unit patients is as high as 30%, And such patients are at increased risk of experiencing in-hospital Complications, compared to patients without diabetes.

Infective complications may be reduced with lower blood glucose concentrations Moreover, in critically ill patients without diabetes, Hyperglycemia is associated with increased mortality, risk of infection, Kidney injury and cardiovascular complications.

Moreover, diabetes is a major risk factor for both Acute Kidney Injury and sepsis.

Sepsis also is a major cause of Acute Kidney Injury, which develops in one-fourth of all patients with sepsis and half of patients with bacteremia or shock .

Sepsis-related Acute Kidney Injury is associated with high mortality rates of up to 70%.

ELIGIBILITY:
Inclusion Criteria:

patients admitted to ICU for any reason and devoloped sepsis either on admission or later during thier hospital stay. patients having Criteria of sepsis or septic shock as defined by 3rd consensus guidelines (sepsis 3) ,2016

Exclusion Criteria:

Previous history of pulmonary problem . Previous history of cardiac disease. Previous history of Autoimmune disease immunocompromised patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted to ICU and devoloped sepsis or septic shock (even on admission or later-on ) as defined by 3rd consensus guidelines (sepsis 3) ,2016 patients then devided into 3 groups : Group 1: patients with Diabetes Mellitus (type 1or type 2). Group 2: patients with in-hospital hyperglycemia(not known to be diabetic). Group 3 : Normglycemic patients (without past or present history of DM ).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
detect the most common organism causing sepsis in ICU . | 20 days
  applying culture and sensitivity tests for patients developed sepsis on admission and follow up will direct us to the proper treatment protocol for all patients.

SECONDARY OUTCOMES:
incidence of sepsis in diabetics versus non diabetics in ICU. | 15 days
  Asses the effect of hyperglycemia on sepsis outcomes.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vincent JL, Marshall JC, Namendys-Silva SA, Francois B, Martin-Loeches I, Lipman J, Reinhart K, Antonelli M, Pickkers P, Njimi H, Jimenez E, Sakr Y; ICON investigators. Assessment of the worldwide burden of critical illness: the intensive care over nations (ICON) audit. Lancet Respir Med. 2014 May;2(5):380-6. doi: 10.1016/S2213-2600(14)70061-X. Epub 2014 Apr 14. PMID 24740011
- [Background] Fleischmann C, Scherag A, Adhikari NK, Hartog CS, Tsaganos T, Schlattmann P, Angus DC, Reinhart K; International Forum of Acute Care Trialists. Assessment of Global Incidence and Mortality of Hospital-treated Sepsis. Current Estimates and Limitations. Am J Respir Crit Care Med. 2016 Feb 1;193(3):259-72. doi: 10.1164/rccm.201504-0781OC. PMID 26414292
- [Background] Jawad I, Luksic I, Rafnsson SB. Assessing available information on the burden of sepsis: global estimates of incidence, prevalence and mortality. J Glob Health. 2012 Jun;2(1):010404. doi: 10.7189/jogh.02.010404. PMID 23198133
- [Background] SepNet Critical Care Trials Group. Incidence of severe sepsis and septic shock in German intensive care units: the prospective, multicentre INSEP study. Intensive Care Med. 2016 Dec;42(12):1980-1989. doi: 10.1007/s00134-016-4504-3. Epub 2016 Sep 29. PMID 27686355
- [Background] Iwashyna TJ, Ely EW, Smith DM, Langa KM. Long-term cognitive impairment and functional disability among survivors of severe sepsis. JAMA. 2010 Oct 27;304(16):1787-94. doi: 10.1001/jama.2010.1553. PMID 20978258
- [Background] Stegenga ME, Vincent JL, Vail GM, Xie J, Haney DJ, Williams MD, Bernard GR, van der Poll T. Diabetes does not alter mortality or hemostatic and inflammatory responses in patients with severe sepsis. Crit Care Med. 2010 Feb;38(2):539-45. doi: 10.1097/CCM.0b013e3181c02726. PMID 19851093
- [Background] Koh GC, Peacock SJ, van der Poll T, Wiersinga WJ. The impact of diabetes on the pathogenesis of sepsis. Eur J Clin Microbiol Infect Dis. 2012 Apr;31(4):379-88. doi: 10.1007/s10096-011-1337-4. Epub 2011 Jul 30. PMID 21805196
- [Background] Bertoni AG, Saydah S, Brancati FL. Diabetes and the risk of infection-related mortality in the U.S. Diabetes Care. 2001 Jun;24(6):1044-9. doi: 10.2337/diacare.24.6.1044. PMID 11375368
- [Background] Luethi N, Cioccari L, Eastwood G, Biesenbach P, Morgan R, Sprogis S, Young H, Peck L, Knee Chong C, Moore S, Moon K, Ekinci EI, Deane AM, Bellomo R, Martensson J. Hospital-acquired complications in intensive care unit patients with diabetes: A before-and-after study of a conventional versus liberal glucose control protocol. Acta Anaesthesiol Scand. 2019 Jul;63(6):761-768. doi: 10.1111/aas.13354. Epub 2019 Mar 18. PMID 30882892
- [Background] Donati A, Damiani E, Domizi R, Botticelli L, Castagnani R, Gabbanelli V, Nataloni S, Carsetti A, Scorcella C, Adrario E, Pelaia P, Preiser JC. Glycaemic variability, infections and mortality in a medical-surgical intensive care unit. Crit Care Resusc. 2014 Mar;16(1):13-23. PMID 24588431
- [Background] Umpierrez G, Cardona S, Pasquel F, Jacobs S, Peng L, Unigwe M, Newton CA, Smiley-Byrd D, Vellanki P, Halkos M, Puskas JD, Guyton RA, Thourani VH. Randomized Controlled Trial of Intensive Versus Conservative Glucose Control in Patients Undergoing Coronary Artery Bypass Graft Surgery: GLUCO-CABG Trial. Diabetes Care. 2015 Sep;38(9):1665-72. doi: 10.2337/dc15-0303. Epub 2015 Jul 15. PMID 26180108
- [Background] de Boer IH, Rue TC, Hall YN, Heagerty PJ, Weiss NS, Himmelfarb J. Temporal trends in the prevalence of diabetic kidney disease in the United States. JAMA. 2011 Jun 22;305(24):2532-9. doi: 10.1001/jama.2011.861. PMID 21693741
- [Background] Venot M, Weis L, Clec'h C, Darmon M, Allaouchiche B, Goldgran-Toledano D, Garrouste-Orgeas M, Adrie C, Timsit JF, Azoulay E. Acute Kidney Injury in Severe Sepsis and Septic Shock in Patients with and without Diabetes Mellitus: A Multicenter Study. PLoS One. 2015 May 28;10(5):e0127411. doi: 10.1371/journal.pone.0127411. eCollection 2015. PMID 26020231
- [Background] Shankar-Hari M, Phillips GS, Levy ML, Seymour CW, Liu VX, Deutschman CS, Angus DC, Rubenfeld GD, Singer M; Sepsis Definitions Task Force. Developing a New Definition and Assessing New Clinical Criteria for Septic Shock: For the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):775-87. doi: 10.1001/jama.2016.0289. PMID 26903336